CLINICAL TRIAL: NCT05956379
Title: Chronic Hepatitis B Patients With Concurrent MAFLD: Cohort Study and Exercise Intervention.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202212084RINC
Record Dates: First submitted 2023-06-13; First posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-06

CONDITIONS: Chronic Hepatitis B; Non-alcoholic Fatty Liver Disease
Keywords: Metabolic syndrome; Exercise intervention; Fatty liver; Chronic Hepatitis B; Gut microbiota
MeSH Terms: conditions — Hepatitis B, Chronic; Non-alcoholic Fatty Liver Disease; Metabolic Syndrome; Fatty Liver | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): Physical therapists will provide personalized aerobic exercise program prescriptions in the preparatory period based on the results of exercise-related assessments, and the training intensity is based on the results of the maximum exercise test, with moderate intensity for 24 weeks, >=3 cardio workouts per week.
  Interventions: Other: exercise
- Control group (No Intervention): No change in exercise habits and maintaining baseline physical activity.

INTERVENTIONS:
Other: exercise — Physical therapists will provide personalized aerobic exercise program prescriptions in the preparatory period based on the results of exercise-related assessments, and the training intensity is based on the results of the maximum exercise test, with moderate intensity for 24 weeks, >=3 cardio workouts per week. The form of aerobic exercise can be carried out in the form of treadmill walking, walking, jogging, cycling, aerobic dance, ball games, swimming, rope skipping, stepping exercises, etc. When the exercise reaches the target intensity, we will adjust the training intensity process according to personal ability. The physical therapist will again adjust the content of the aerobic exercise program at week 12 based on the reassessment of the exercise capacity.
  Arms: Exercise group

SUMMARY:
In Taiwan, HBV infection is endemic in the adult population. With the westernization of eating habit and lifestyle, metabolic syndrome and related non-alcoholic fatty liver diseases (NAFLD, newly proposed as metabolic dysfunction associated fatty liver diseases, MAFLD) has become another important health issue. It is therefore common to encounter subjects with concurrent MAFLD and HBV infection in HBV endemic countries. This project will study the clinical data of patients with concurrent MAFLD and HBV, and aim to explore the impact of exercise intervention on the hepatic fatty infiltration, alteration of gut microbiota and HBV replication status in this group of patients. The research strategies will include (1) improving fatty liver and metabolic syndrome in subjects with concurrent MAFLD and HBV; and (2) exploring the changes of HBV replication and intestinal microflora in patients with concurrent HBV and MAFLD after exercise intervention.

DETAILED DESCRIPTION:
The investigators will first collect and analyze clinical data of patients with concurrent MAFLD and HBV in a retrospective cohort in NTUH. The investigators aim to clarify the interactions of MAFLD and HBV based on different HBV-related liver disease stage and different metabolic derangement.

Second, using the well-established platform for the detection and staging of fatty liver at NTUH, the investigators plan to enroll 100 patients with concurrent HBV and MAFLD. The investigators will collect all basic information including intrahepatic fat and fibrosis severity, and randomize them to the exercise intervention group (n = 50) and the observation group (n = 50) after conditional screening. After 6-month of exercise intervention, the investigators will analyze the effect of exercise on intrahepatic fat (main parameter: 10% reduction in intrahepatic fat; 30% achieved in the exercise intervention group; 5% achieved in the control group) and analyze the influence of co-existing HBV on the change of hepatic steatosis.

Description of the prospective randomized exercise intervention studies

1. Enrolment of 100 patients with concurrent chronic HBV infection and MAFLD
2. Collection of baseline data: Clinical parameters, virologic parameters, metabolic and MAFLD parameters, nutritional and exercise fitness data, and liver steatosis/fibrosis data
3. Randomization: Randomization into exercise (Group I) versus non-exercise group (Group II) will be conducted with the help of random number table.
4. 24-week exercise intervention
5. 12-week post-exercise follow-up period
6. Collection of final data, statistical analyses and paper preparation

II-1: Enrolment of subjects:

Patients from NTUH with the diagnosis of chronic HBV infection will be screened for the presence of MAFLD at the out-patient clinics. Treatment naïve patients found to have co-existing MAFLD and willing to join the active exercise program will be invited to join the study by the clinical physicians after thorough evaluation. Patients with age less than 18 years, concurrent HCV or HIV co-infection will be excluded.

CHB patients fulfilling reimbursement criteria for the treatment of HBAg-positive or -negative CHB, or advanced fibrosis/cirrhosis will not be enrolled since the virologic profiles under NUC therapy would not likely to be affected by the change of hepatic steatosis through exercise intervention.

Assessment of HBV replication status and liver disease severity: The clinical phenotype of HBV infection will be determined by liver function test (serum ALT level) and platelet count number, abdominal ultrasonography, FibroScan™, along with serum HBeAg and HBV DNA level. At enrolment, the patients will be categorized into HBeAg positive chronic HBV infection (immune tolerance phase), HBeAg positive chronic hepatitis B (immune clearance phase), HBeAg negative chronic HBV infection (low replication phase), and HBeAg negative chronic hepatitis B (reactivation phase). The stage of liver fibrosis will determined by FIB-4, FibroScan™and MR elastography (MRE).

Diagnosis and assessment of MAFLD: The diagnosis of MAFLD will be made if the patient has evidence of hepatic steatosis by both abdominal ultrasonography and FibroScan™, along with one of the three criteria, namely overweight/obesity, presence of type 2 diabetes mellitus (DM), and at least two metabolic risk abnormalities. Then the degree of hepatic steatosis and fibrosis will be semi-quantitatively assessed by FibroScan™. In this proposal, the investigators will for the first time adopt MR PDFF and MR elastography (MRE) to accurately assess the degree of steatosis and the stage of fibrosis in each enrolled subject before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years of age
* Either gender
* HBV treatment naïve
* Capable of taking exercise
* HBsAg positivity for >6 months
* Evidence of fatty liver in both abdominal ultrasonography and Fibroscan™(CAP>215)

Exclusion Criteria:

* Age >70 years of age
* Evidence of liver cirrhosis
* Patients fulfilling reimbursement criteria for HBV treatment
* Evidence of severe cardiopulmonary diseases
* Evidence of serious hip or knee problems, incapable of taking exercise
* Evidence of liver decompensation
* Evidence of active HCV (positive for serum HCV RNA) or HIV infection (positive for anti-HCV)
* Clinical diagnosis of Alzheimer's Disease
* Thyroid disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Change of hepatic steatosis after 6-month exercise intervention by MRI-PDFF | 24 weeks
  We will measure change of hepatic steatosis at week 24 in comparison to baseline steatosis by MRI-PDFF. Reduction of hepatic steatosis by >=10% will be defined as responder.

OTHER OUTCOMES:
Exploratory outcomes | 24 weeks
  1. Dynamics of HBV profiles after exercise
  2. Impact of diminishing hepatic steatosis on the evolution of liver fibrosis
  3. Impact of diminishing hepatic steatosis on the profiles of HBV replication

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Jen Liu, Professor, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Zhongzheng Dist., Taiwan

IPD SHARING:
Plan to Share IPD: No